CLINICAL TRIAL: NCT06682234
Title: A Phase 2, Single-Arm Study of Obeldesivir for Postexposure Prophylaxis of Filovirus Diseases
Brief Title: Study of Obeldesivir as Postexposure Prophylaxis for Filovirus Diseases Virus Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GS-US-719-7450
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Filovirus Disease; Postexposure Prophylaxis for Filovirus Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Obeldesivir (ODV) (Experimental): Participants will receive ODV for 10 days
  Interventions: Drug: obeldesivir

INTERVENTIONS:
Drug: obeldesivir — Tablets administered orally
  Other Names: GS-5245

SUMMARY:
The goal of this clinical study is to learn more about the study drug, obeldesivir (ODV), and how safe and effective it is preventing Filovirus disease in participants with known or suspected exposure to Filovirus disease.

The primary objective is to evaluate the safety and tolerability of ODV for Ebola virus (EBOV), Sudan virus (SUDV), and MARV postexposure prophylaxis (PEP).

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and give written informed consent and comply with treatment and follow up.
* Individuals who are of childbearing potential and engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception
* Known or suspected high-risk exposure to Ebola virus (EBOV), Sudan virus (SUDV), or Marburg virus (MARV) within 21 days of Day 1. High-risk exposure may include the following:

  1. Direct contact with bodily fluids from a confirmed case.
  2. Needle stick injury with a needle potentially contaminated with virus.
  3. Prolonged exposure to an individual with EBOV, SUDV, or MARV infection or disease without (adequate) personal protective equipment.

Key Exclusion Criteria:

* Individuals with plans to breastfeed during the study period and 21 days following the last dose of study intervention. World Health Organization guidance on breastfeeding should be followed.
* Known hypersensitivity to the study intervention, its metabolites, or formulation excipient.
* Known EBOV, SUDV, or MARV reverse transcriptase-polymerase chain reaction (RT-PCR) positivity or symptomatic filovirus disease as attributed by the investigator.
* Known moderate or severe renal impairment or known estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m^2.
* Decompensated cirrhosis (Child-Pugh Class C), acute liver injury/failure (eg, new onset [< 2 weeks] of easy bruising, jaundice, ascites, hepatic encephalopathy, asterixis), and/or known alanine aminotransferase ≥5 × upper limit of normal.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Serious Adverse Events (SAEs) | First dose date up to 29 Days

SECONDARY OUTCOMES:
Proportion of Participants with Symptomatic Filovirus Disease by Day 29 | Up to 29 Days
Proportion of Participants with Polymerase Chain Reaction (PCR)-Confirmed Filovirus Disease Infections by Day 29 | Up to 29 Days
Proportion of Participants with All-Cause Death by Day 29 | Up to 29 Days

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06682234